CLINICAL TRIAL: NCT03343431
Title: A Maternal Short Course of Tenofovir Disoproxil Fumarate and Infant Vaccine to Prevent Mother-to-child Transmission of Hepatitis B Virus
Brief Title: Antiviral Prophylaxis and Infant Vaccination to Prevent Perinatal Hepatitis B Infection
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Institut de Recherche pour le Developpement (Other Government)
Collaborators: Chiang Mai University (Other); Ministry of Health, Thailand (Other Government); Ministry of Health, Lao PDR (Unknown)
Responsible Party: Principal Investigator, GONZAGUE JOURDAIN, Researcher, Institut de Recherche pour le Developpement
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: iTAP-2
Record Dates: First submitted 2017-11-06; First posted 2017-11-17 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Hepatitis B; Pregnancy
Keywords: Hepatitis B; Hepatitis B eAg; Pregnancy
MeSH Terms: conditions — Hepatitis B | interventions — Tenofovir

STUDY DESIGN:
Intervention Model Description: All participants receive the intervention
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Anti-HBV antiviral prophylaxis — Tenofovir disoproxil fumarate (TDF), one 300 mg tablet once a day from 28 weeks' gestation through two months postpartum
  Other Names: tenofovir disoproxil fumarate

SUMMARY:
Most new hepatitis B virus (HBV) infections are acquired perinatally. In this study, pregnant women with HBsAg and HBeAg will receive tenofovir disoproxil fumarate during the last trimester of pregnancy and for two months following delivery. Their infants will receive hepatitis B (HB) immunization, starting with a first dose soon after birth. We hypothesize that the risk of mother-to-child transmission of HBV will be lower than 2%. The results of the study will help define policy to manage HBV infected pregnant women to prevent perinatal transmission.

DETAILED DESCRIPTION:
This is a prospective multi-center, multi-country (Thailand and Lao PDR), open-label, single arm clinical trial in HBsAg and HBeAg positive pregnant women (from 28 weeks until one year postpartum) and their infants (until 18 months of age). Pregnant women with HBsAg and HBeAg will receive tenofovir disoproxil fumarate 300 mg once daily from 28 weeks of pregnancy until two months postpartum. Their infants will receive hepatitis B (HB) immunization, starting with the first dose soon after birth.

The study aims to show that substituting maternal antiviral treatment for infant HBIg can be favorably considered in settings where HBIg plus vaccine has been used as well as in settings where only vaccine is used. A significant improvement over the standard HBIg + vaccine strategy would be that adding an antiviral strategy results in less than 2% transmission. A total of 499 women and their infants will be enrolled in public hospitals in Thailand and Lao PDR.

The study will be monitored by a Data and Safety Monitoring Board (DSMB) at least annually.

ELIGIBILITY:
Inclusion Criteria:

* Pregnancy
* Age ≥18 years
* Negative HIV antibody test during current pregnancy
* Positive HBsAg test during current pregnancy
* Positive HBeAg using a rapid test during current pregnancy
* Absence of clinical symptoms of liver disease
* Gestational age of 28 weeks (+/- 7 days) based on the obstetrician judgment guided by the review of the date of last menstruation period.
* Willing and able to provide written informed consent
* Agreeing to bring her infants(s) at the planned study visits at one of the study site until the last visit (18 months after birth) and to inform the site investigators if plans to move to another place and not be able to return to the clinic
* Understand the need for adequate infant immunization for her infant(s) and accept that blood draws will be performed to determine the infant HBV infection status

Exclusion Criteria:

* Receipt of anti-HBV antivirals at any time during the last 9 months
* Known liver cirrhosis or evidence of hepatocellular carcinoma
* Creatinine clearance <50 ml/min, calculated using the Cockcroft-Gault formula
* Confirmed dipstick proteinuria >1+ (>30 mg/dL) or normoglycemic glycosuria
* Evidence of pre-existing fetal anomalies incompatible with life
* Any concomitant condition or treatment that, in the view of the clinical site investigator, would contraindicate participation or compromise adherence to treatment and satisfactory follow up in the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Pregnant women
Enrollment: 504 (Actual)
Dates: Start 2018-08-02 (Actual); Primary Completion 2023-05-13 (Actual); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Infant hepatitis B infection status | Six months of age
  HBsAg positive confirmed by PCR detection of HBV DNA.

SECONDARY OUTCOMES:
Maternal HBV DNA changes | From enrollment until end of study treatment scheduled 2 months after delivery
  Description of the effect of tenofovir disoproxil fumarate on maternal HBV DNA levels
Infant levels of anti-HBs antibodies | At 1, 2, 4, 6, and 12 months of age
  Levels of anti-HBs antibodies in infants in the absence of HBIg administration at birth
HBV infection status in all infants regardless of maternal response to study treatment | At 6 months of age
  HBsAg positive confirmed by PCR detection of HBV DNA in all infants, i.e. including those born to women with unsatisfactory virological response to study treatment
Serious adverse events | From enrollment until 12 months postpartum
  Occurrence of maternal serious adverse events (ICH SAEs) including DAIDS grade 4 signs and symptoms regardless of their relatedness to the study treatment
Serious adverse events | From birth until 12 months of age
  Occurrence of infant serious adverse events (ICH SAEs) including DAIDS grade 4 signs and symptoms regardless of their relatedness to the study treatment
Preterm live births | Delivery
  Proportion of neonates born alive before 37 weeks of pregnancy
Low birth weight | Delivery
  Proportion of neonates born alive with birth weight of 2,499 g or less, regardless of gestational age
Active or previous transient infection in children | At 18 months of age
  Detection of anti-HBc antibodies among all infants

CONTACTS AND LOCATIONS:
Overall Officials: Gonzague Jourdain, MD, PhD, Principal Investigator — Chiang Mai University
Locations (20):
- Laos (8):
  - Champasak Hospital, Champasak
  - Luang Prabang Provincial Hospital, Luang Prabang
  - Sayaboury Hospital, Sainyabuli
  - Savannakhet Provincial hospital, Savannakhet
  - 103 Hospital, Vientiane
  - Mahosot Hospital, Vientiane
  - Mother and Newborn Hospital, Vientiane
  - Setthathirath Hospital, Vientiane
- Thailand (12):
  - Chiang Kham Hospital, Chiang Kham, Changwat Phayao
  - Nopparat Rajathanee Hospital, Bangkok
  - Prapokklao Hospital, Chanthaburi
  - Health Promotion Center Region 1, Chiang Mai
  - Nakornping Hospital, Chiang Mai
  - Chiangrai Prachanukroh Hospital, Chiang Rai
  - Chonburi Hospital, Chon Buri
  - Banglamung Hospital, Chon Buri
  - Lampang Hospital, Lampang
  - Lamphun Hospital, Lamphun
  - Samutprakarn Hospital, Mueang Samut Prakan
  - Samutsakhon Hospital, Samut Sakhon

IPD SHARING:
Plan to Share IPD: Yes
We are willing to share our data to answer important research questions requiring large datasets, after completion of the original research plan and substudies. Data-sharing agreements will include: an approval of the research plan by appropriate ethics committees, a commitment to using data for research purposes only and to securing the data or/and the samples using appropriate methods. Data used for publications will be released in a timely manner. De-identified study data will be accessible through the Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) Data and Specimen Hub or DASH (dash.nichd.nih.gov/).
  However, as of May 25, 2025, the DASH website will be unable to support new submissions for the next several months. The PI will submit the data when new submissions are open.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: At the same time as related publications
Access Criteria: See Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) Data and Specimen Hub or DASH
URL: https://dash.nichd.nih.gov

DOCUMENTS (3):
  • Study Protocol (2020-12-02): https://cdn.clinicaltrials.gov/large-docs/31/NCT03343431/Prot_006.pdf
  • Statistical Analysis Plan (2023-11-30): https://cdn.clinicaltrials.gov/large-docs/31/NCT03343431/SAP_005.pdf
  • Informed Consent Form (2020-01-15): https://cdn.clinicaltrials.gov/large-docs/31/NCT03343431/ICF_007.pdf